CLINICAL TRIAL: NCT04344756
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients CORIMUNO-COAG Trial
Brief Title: Trial Evaluating Efficacy and Safety of Anticoagulation in Patients With COVID-19 Infection, Nested in the Corimmuno-19 Cohort
Acronym: CORIMMUNO-COAG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200389-6
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID19 Pneumonia
MeSH Terms: interventions — Tinzaparin; Heparin

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 2 parallels arms, 1:1, stratified on disease severity (ventilation or not)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Coagulation (Experimental)
  Interventions: Drug: Tinzaparin or unfractionated heparin
- Standard of Care (No Intervention): Control patients will receive the best standard of care and a subcutaneous preventive anticoagulation for at least 14 days with enoxaparin 4000 IU/24h, tinzaparin 3500 IU/24h or dalteparin 5000 IU/24h if creatinine clearance (Cockcroft) ≥ 30mL/min or unfractionated heparin 5000 IU/12h if creatinine clearance < 30mL/min.

INTERVENTIONS:
Drug: Tinzaparin or unfractionated heparin — Tinzaparin INNOHEP ® 175 IU/kg/24h for 14 days if creatinine clearance Cockcroft ≥ 20mL/min, Otherwise unfractionated heparin (Calciparine®, Héparine Sodique Choay®) subcutaneously or intravenous with an anti-Xa target between 0.5 and 0.7 IU/mL for 14 days
  Arms: Active Coagulation

SUMMARY:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) and causes substantial morbidity and mortality. There is currently no vaccine to prevent Covid-19 or infection with SARS-CoV-2 or therapeutic agent to treat COVID-19.

This protocol CORIMUNO19-COAG will evaluate the efficacy and safety of active anticoagulation using heparin: Tinzaparin (INNOHEP®) or unfractionated heparin (Calciparine®, Héparine Sodique Choay®) in COVID-19 patients hospitalized in conventional or intensive care units.

It will use a phase 2 randomized open-label multicentre clinical trial, where patients will be randomly allocated to anticoagulation versus Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

1. group 1 : patients not requiring ICU at admission with mild disease to severe pneumopathy according to The Who Criteria of severity of COVID pneumopathy, and with symptom onset before 14 days, with need for oxygen but No non-invasive ventilation (NIV) or High flow
2. group 2 :

   * Respiratory failure AND requiring mechanical ventilation
   * WHO progression scale ≥ 6
   * No do-not-resuscitate order (DNR order)

Exclusion Criteria:

* Patients with contraindications to anticoagulation

  1. Congenital hemorrhagic disorders
  2. Hypersensitivity to tinzaparin or UHF or to any of the excipients
  3. Current or history of immune-mediated heparin-induced thrombocytopenia
  4. Active major haemorrhage or conditions predisposing to major haemorrhage. Major haemorrhage is defined as fulfilling any one of these three criteria: a) occurs in a critical area or organ (e.g. intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, intra-uterine or intramuscular with compartment syndrome), b) causes a fall in haemoglobin level of 20 g/L (1.24 mmol/L) or more, or c) leads to transfusion of 2 or more units of whole blood or red blood cells.
  5. Septic endocarditis
* Patients with need for anticoagulant therapy. For example: atrial fibrillation, venous thromboembolism, mechanical valve, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Survival without ventilation (VNI or mechanical ventilation) | day 14
  group 1
ventilator free survival | day 28
  group 2

SECONDARY OUTCOMES:
World Health Organisation(WHO) progression scale ≤5 | day 4
  range from 0 (healthy) to 10 (death) values below or equal to 5 correspond to the absence of any oxygen supply beside nasal or facial mask
World Health Organisation(WHO) progression scale | day 4, 7 and 14
  range from 0 (healthy) to 10 (death)
overall survival | day 14, 28 and 90
Length of hospital stay | day 28
Length of ICU stay | day 28
time to oxygenation supply independency | day 28
time to ventilator (non invasive or invasive) | day 28
rate of acute kidney injury | day 28
  according to Acute Kidney Injury (AKIN) classification system
time to Renal Replacement Therapy (RRT) initiation | day 28
rate of clinically overt pulmonary embolism or proximal deep vein thrombosis | day 14 and day 90
  confirmed by objective testing
Rate of clinically overt arterial thrombosis | day 14 and day 90
  confirmed by objective testing
Rate of unscheduled central venous catheter replacement for catheter dysfunction | day 28
Rate of central venous catheter-related deep vein thrombosis (CVC-DVT) | day 28
  as a thrombus extending from the catheter into the lumen of the deep vein where the catheter is inserted diagnosed with radiologic imaging in case of a clinical suspicion of upper/lower limb DVT or pulmonary embolism or compulsory catheter removal
Rate of unscheduled indwelling arterial catheter replacement for catheter dysfunction | day 28
Rate of acute clotting leading to the replacement the renal replacement therapy circuit stratified by regional citrate anticoagulation or not | day 28
Time to acute clot formation within the oxygenator (acute oxygenator thrombosis, AOT) leading to the exchange of an extracorporeal membrane oxygenation (ECMO) system | day 28
Time to acute clot formation within the pump head (pump head thrombosis, PHT) leading to the exchange of an extracorporeal membrane oxygenation (ECMO) system | day 28
Incidence of adverse events | day 28

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Réanimation hôpital Louis Mourier, Colombes, Hauts De Seine
  - réanimation hôpital Cochin, Paris
  - Médecine vasculaire, Hôpital Européen Georges Pompidou, Paris

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773